CLINICAL TRIAL: NCT00311480
Title: A Phase II, Randomized, Controlled, Observer-Blind, Multi-Center Study to Evaluate Safety and Immunogenicity of Two Doses, Administered Three Weeks Apart, of Two (Surface Antigen Adjuvanted With MF59C.1) Influenza Vaccines Containing 7.5 mg or 15 mg of H5N1 Influenza Antigen, in Non-Elderly Adult and Elderly Subjects
Brief Title: Safety and Immunogenicity of Two Doses, Administered Three Weeks Apart, of Two(Surface Antigen Adjuvanted With MF59C.1) Influenza Vaccines in Non-Elderly Adult and Elderly Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: V87P1; Eudract:2005-005871-14
Record Dates: First submitted 2006-04-04; First posted 2006-04-06 (Estimated); Last update posted 2007-03-13 (Estimated); Status verified 2007-03

CONDITIONS: Pandemic Influenza Disease
Keywords: influenza; pandemic influenza; influenza vaccine; adjuvanted influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — MF59 oil emulsion

INTERVENTIONS:
Biological: Influenza vaccine surface antigen adjuvanted with MF59

SUMMARY:
The present study aims to evaluate safety and immunogenicity of two doses, administered three weeks apart, of two influenza vaccines containing 7.5 micrograms or 15 micrograms of H5N1 influenza antigen, in non-elderly adult and elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers 18 years of age or older

Exclusion Criteria:

* any auto-immune disease or other serious acute, chronic or progressive disease
* hypersensitivity to eggs, chicken protein, chicken feathers, influenza viral protein, neomycin or polymyxin or any other component of the vaccine.
* history of neurological symptoms or signs, or anaphylactic shock following administration of any vaccine.
* within the past 7 days, they have experienced: any acute disease, infections requiring systemic antibiotic or antiviral therapy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 520
Dates: Start 2006-03

PRIMARY OUTCOMES:
CPMP criteria for evaluation of flu vaccines e.g. Seroprotection, GMT's and Seroconversion rate at day 0 and day 22 and day 43 following vaccination

SECONDARY OUTCOMES:
Solicited Local and Systemic Reactions Within 6 Days Following Each Vaccination And Adverse Events Thought the Study.

CONTACTS AND LOCATIONS:
Overall Officials: Drug Information Services, Principal Investigator — Novartis Vaccines & Diagnostics
Locations (4):
- Italy (4):
  - G. D'Annunzio University, Chieti
  - Department of Health Sciences, Genoa
  - ASL Lanciano-Vasto, Lanciano
  - University Hospital of Siena, Siena

REFERENCES:
- [Derived] Banzhoff A, Gasparini R, Laghi-Pasini F, Staniscia T, Durando P, Montomoli E, Capecchi PL, di Giovanni P, Sticchi L, Gentile C, Hilbert A, Brauer V, Tilman S, Podda A. MF59-adjuvanted H5N1 vaccine induces immunologic memory and heterotypic antibody responses in non-elderly and elderly adults. PLoS One. 2009;4(2):e4384. doi: 10.1371/journal.pone.0004384. Epub 2009 Feb 6. PMID 19197383